CLINICAL TRIAL: NCT00526383
Title: Do Antidepressants Induce Metabolic Syndromes
Brief Title: Do Antidepressants Induce Metabolic Syndromes METADAP Study
Acronym: METADAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P060219
Record Dates: First submitted 2007-09-05; First posted 2007-09-10 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2007-09

CONDITIONS: Major Depressive Disorder
Keywords: Major depressive disorder; Antidepressants; Weight gain; Metabolic syndromes
MeSH Terms: conditions — Depressive Disorder, Major; Weight Gain; Metabolic Syndrome | interventions — Antidepressive Agents, Tricyclic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): antidepressant versus medical dispositive
  Interventions: Drug: Tricyclic antidepressants
- B (Placebo Comparator)
  Interventions: Drug: Tricyclic antidepressants

INTERVENTIONS:
Drug: Tricyclic antidepressants — antidepressant version medical dispositive
  Other Names: antidepressant version medical dispositive

SUMMARY:
Since antidepressants and antipsychotics have common receptorial mechanisms of action (H1 antagonism, 5HT2 antagonism), the impact of antidepressants in terms of metabolic syndromes is a matter of concern.

The main objective of this study is to assess the differential impact of antidepressants in terms of weight gain and metabolic syndromes.

DETAILED DESCRIPTION:
Since antidepressants and antipsychotics have common receptorial mechanisms of action (H1 antagonism, 5HT2 antagonism), the impact of antidepressants in terms of metabolic syndromes is a matter of concern.

The main objective of this study is to assess the differential impact of antidepressants in terms of weight gain and metabolic syndromes.

Prospective 6-month naturalistic cohort study, comparing 4 classes of antidepressants (SSRIs, SNRIs, TCAs and others) to a control group (ECT and r-TMS), in 600 patients with a major depressive disorder requiring the beginning of either antidepressant or ECT/r-TMS treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age : 18-70
* Current major depressive episode (Major depressive disorder) based on the MINI interview
* HAM-D >18
* Requiring either antidepressant treatment, either ECT or r-TMS (as assessed by the clinician)
* Signed informed consent

Exclusion Criteria:

* Bipolar disorder (DSM-IV), Psychotic disorder (DSM-IV), Substance abuse or dependence (DSM-IV)
* Normothymic treatment
* Antipsychotic treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 624 (Actual)
Dates: Start 2007-11; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Definition criteria of the metabolic syndromes: Weight and waist circumference Systolic and diastolic blood pressure Glycemia Triglyceridemia Cholesterolemia Insulinemia | at Months 0, 1, 3, 6

SECONDARY OUTCOMES:
Antidepressant efficacy (HAM-D, quickIDS-C, quickIDS-SR, CGI) | at Months 0, 1, 3, 6

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle CORRUBLE, MD PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Assistance Publique hopital Bicêtre, Paris, France

REFERENCES:
- [Derived] Chappell K, Ait Tayeb AEK, Colle R, Bouligand J, El-Asmar K, Gressier F, Trabado S, David DJ, Feve B, Becquemont L, Corruble E, Verstuyft C. The association of ARRB1 polymorphisms with response to antidepressant treatment in depressed patients. Front Pharmacol. 2022 Oct 26;13:974570. doi: 10.3389/fphar.2022.974570. eCollection 2022. PMID 36386175
- [Derived] Chappell K, Colle R, Ait Tayeb AEK, Bouligand J, El-Asmar K, Deflesselle E, Feve B, Becquemont L, Corruble E, Verstuyft C. The ERICH3 rs11580409 polymorphism is associated with 6-month antidepressant response in depressed patients. Prog Neuropsychopharmacol Biol Psychiatry. 2022 Dec 20;119:110608. doi: 10.1016/j.pnpbp.2022.110608. Epub 2022 Jul 22. PMID 35878676
- [Derived] Loeb E, Becquemont L, Corruble E. Is the decrease in NOx due to a lack of substrate or a NOS inhibition in patients with major depression? : Commentary on Hess et al. 2017. Psychopharmacology (Berl). 2021 Feb;238(2):613-614. doi: 10.1007/s00213-020-05747-x. Epub 2021 Jan 9. No abstract available. PMID 33420804
- [Derived] Loeb E, El Asmar K, Trabado S, Gressier F, Colle R, Rigal A, Martin S, Verstuyft C, Feve B, Chanson P, Becquemont L, Corruble E. Nitric Oxide Synthase activity in major depressive episodes before and after antidepressant treatment: Results of a large case-control treatment study. Psychol Med. 2022 Jan;52(1):80-89. doi: 10.1017/S0033291720001749. Epub 2020 Jun 11. PMID 32524920